CLINICAL TRIAL: NCT00383669
Title: Trial of Vitamins in HIV Progression and Transmission (A Trial of Vitamins and HAART in HIV Disease Progression)
Brief Title: A Trial of Vitamins and HAART in HIV Disease Progression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Wafaie Fawzi, Chair, Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HD32257-01; P12981-101
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: HIV; AIDS; Disease Progression; Multivitamins; Anti-Retroviral Therapy; HAART; Tanzania; Africa
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Disease Progression | interventions — Geritol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple RDA multivitamins (Active Comparator): Multivitamins (including B, C, and E)
  Interventions: Dietary Supplement: Multivitamins (including B, C and E)
- Single RDA Multivitamins (Active Comparator): Multivitamins (including B, C, and E)
  Interventions: Dietary Supplement: Multivitamins B, C and E

INTERVENTIONS:
Dietary Supplement: Multivitamins (including B, C and E) — One daily oral dose of 20 mg B1, 20 mg B2, 25 mg B6, 100 mg niacin, 50 μg B12, 0.8 mg folic acid, 500 mg C, and 30 mg vitamin E taken taken from randomization until the end of follow-up (24-28 months).
  Arms: Multiple RDA multivitamins
Dietary Supplement: Multivitamins B, C and E — One daily oral dose of 1.2 mg vitamin B1, 1.2 mg vitamin B2, 1.3 mg vitamin B6, 15 mg niacin, 2.4 μg vitamin B12, 0.4 mg folic acid, 80 mg vitamin C, and 15 mg vitamin E taken taken from randomization until the end of follow-up (24-28 months).
  Arms: Single RDA Multivitamins

SUMMARY:
This study is a double-blind randomized clinical trial, conducted to examine the effects of multivitamins (including B, C, and E) on HIV disease progression among HIV-positive Tanzanian adult men and women taking highly active anti-retroviral therapy (HAART).

DETAILED DESCRIPTION:
Access to Highly Active Anti-Retroviral Therapy (HAART) for the treatment of HIV in developing regions is limited, but gradually becoming standard of care in some countries. Multivitamin supplements have demonstrated immune-enhancing effects among individuals in pre-HAART HIV disease stages. However, the efficacy and safety of micronutrient supplements need to be documented in the context of HAART. This study is a double-blind randomized clinical trial, conducted to examine the effect of multivitamins (including B, C, and E) on HIV disease progression among individuals taking HAART. Participants are HIV-positive Tanzanian men and women aged 18 years and older, who are initiating HAART at the time of randomization. Eligible individuals are randomized to receive daily oral supplements in one of two intervention groups: a) multivitamins at the single Recommended Dietary Allowance (RDA) level; and b) multivitamins at multiples of the RDA at the same doses used in our previous study "A Trial of Vitamins in HIV Progression and Transmission".

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Men or Women
* 18 Years of Age or older
* Initiating HAART at time of randomization

Exclusion Criteria:

* Pregnant or Lactating Women
* Individuals at pre-HAART disease stages
* BMI less than 16

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4012 (Actual)
Dates: Start 2006-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Development of a new or recurrent disease progression event, including all-cause death. | within 24 months after randomization

SECONDARY OUTCOMES:
Changes in: (a) CD4 cell count, (b) plasma HIV-1 RNA concentration, (c) weight, and (d) alteration to second-line anti-retroviral treatment; and occurrence of (a) adverse events, specifically peripheral neuropathy | within 24 months of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MD,DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Muhimbili University College of Health Sciences, Dar es Salaam, Tanzania

REFERENCES:
- [Derived] Abioye AI, Hughes MD, Sudfeld CR, Noor RA, Isanaka S, Lukmanji Z, Mugusi F, Fawzi WW. Dietary Iron Intake and HIV-Related Outcomes Among Adults Initiating Antiretroviral Therapy in Tanzania. J Acquir Immune Defic Syndr. 2023 Sep 1;94(1):57-65. doi: 10.1097/QAI.0000000000003221. PMID 37199401
- [Derived] Noor RA, Abioye AI, Hertzmark E, Darling AM, Aboud S, Mugusi FM, Sudfeld CR, Spiegelman D, Fawzi WW. Impaired Hematological Status Increases the Risk of Mortality among HIV-Infected Adults Initiating Antiretroviral Therapy in Tanzania. J Nutr. 2020 Sep 1;150(9):2375-2382. doi: 10.1093/jn/nxaa172. PMID 32621487
- [Derived] Abioye AI, Isanaka S, Liu E, Mwiru RS, Noor RA, Spiegelman D, Mugusi F, Fawzi W. Gender differences in diet and nutrition among adults initiating antiretroviral therapy in Dar es Salaam, Tanzania. AIDS Care. 2015;27(6):706-15. doi: 10.1080/09540121.2014.996517. Epub 2015 Jan 6. PMID 25562355
- [Derived] Sudfeld CR, Isanaka S, Mugusi FM, Aboud S, Wang M, Chalamilla GE, Giovannucci EL, Fawzi WW. Weight change at 1 mo of antiretroviral therapy and its association with subsequent mortality, morbidity, and CD4 T cell reconstitution in a Tanzanian HIV-infected adult cohort. Am J Clin Nutr. 2013 Jun;97(6):1278-87. doi: 10.3945/ajcn.112.053728. Epub 2013 May 1. PMID 23636235
- [Derived] Isanaka S, Mugusi F, Hawkins C, Spiegelman D, Okuma J, Aboud S, Guerino C, Fawzi WW. Effect of high-dose vs standard-dose multivitamin supplementation at the initiation of HAART on HIV disease progression and mortality in Tanzania: a randomized controlled trial. JAMA. 2012 Oct 17;308(15):1535-44. doi: 10.1001/jama.2012.13083. PMID 23073950

DOCUMENTS (1):
  • Informed Consent Form (2006-07-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT00383669/ICF_000.pdf